CLINICAL TRIAL: NCT00313560
Title: Phase II Study of Erlotinib (TarcevaTM) Combined With Chemoradiation and Adjuvant Chemotherapy in Patients With Resectable Pancreatic Cancer
Brief Title: ChemoRT With Adjuvant Chemo in Pancreatic Cancer (TARCEVA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0534; R01CA104900 (NIH); P30CA006973 (NIH); NA_00025965 (Other: JHM IRB); JHOC-05080408; GENENTECH-JHOC-J0534; CDR0000465208 (Other: other); NCT00962520 (obsolete NCT alias)
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage I pancreatic cancer; stage II pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Erlotinib and EBRT after pancreatectomy (Experimental): Adjuvant treatment with erlotinib 100 mg plus Capecitabine 800 mg/m2 PO BID (5 days on/ 2 days off regimen) and External Beam Radiation Therapy (EBRT) at doses of 50.4 Gy in 28 fractions after pancreatectomy (Dosing for capecitabine and erlotinib was amended after considering the toxicity profile of the first 6 patients).
  Approximately 4-8 weeks after the conclusion of chemoradiation, it is recommended patients will continue treatment with 4 cycles of gemcitabine 1000 mg/m2 days 1, 8, and 15 every 28 days plus daily erlotinib 100 mg.
  Interventions: Drug: erlotinib hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride — Erlotinib 100 mg PO QD (1 hour prior to Capecitabine) (both given daily without interruption)
  Other Names: Tarceva

SUMMARY:
To seek preliminary evidence of antitumor activity (progression free survival) of Erlotinib in combination with standard adjuvant chemoradiation and chemotherapy in patients with resected adenocarcinoma of the pancreas.

DETAILED DESCRIPTION:
This study is a phase II trial of erlotinib in combination with chemoradiation in patients with stage I/II adenocarcinoma of the pancreas who are candidates for adjuvant chemoradiation.

This study is a phase II trial of erlotinib in combination with chemoradiation in patients with resected stage I/II adenocarcinoma of the pancreas who are candidates for adjuvant chemoradiation. Eligible patients will receive adjuvant treatment with erlotinib 100 mg plus Capecitabine 800 mg/m2 PO BID (5 days on/ 2 days off regimen) and External Beam Radiation Therapy (EBRT) at doses of 50.4 Gy in 28 fractions after pancreatectomy (Dosing for capecitabine and erlotinib was amended after considering the toxicity profile of the first 6 patients). Approximately 4-8 weeks after the conclusion of chemoradiation, it is recommended patients will continue treatment with 4 cycles of gemcitabine 1000 mg/m2 days 1, 8, and 15 every 28 days plus daily erlotinib 100 mg.

Eligible patients will receive adjuvant treatment with erlotinib 100 mg plus Capecitabine 800 mg/m2 PO BID (5 days on/ 2 days off) and External Beam Radiation Therapy (EBRT) to the tumor bed plus adjacent lymph nodes at doses of 50.4 Gy in 28 fractions after surgery. For patients with close or positive margins after resection, they will be able to receive 54.0 Gy over 30 fractions. Approximately 4-8 weeks after the conclusion of chemoradiation, it is recommended patients will continue treatment with 4 cycles of gemcitabine 1000 mg/m2 days 1, 8, and 15 every 28 days plus erlotinib 100 mg/daily.

ELIGIBILITY:
Inclusion criteria

1. Resection of a stage I/II pancreatic adenocarcinoma of the pancreas (R0/R1) and a candidate to receive postoperative adjuvant chemoradiation. R2 (laparoscopic resection) based on the surgeons operative note will be excluded from the study.
2. Aged 18 years or older.
3. ECOG performance status < 1.
4. The effects of Erlotinib and Capecitabine on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
5. Patients must have normal organ and marrow function.
6. Provision of written informed consent
7. Patients must have a working knowledge of English in order to complete the quality of life questionnaires. Patients that do not meet this requirement will be exempt from the QoL assessment, but remain eligible for all other components of the study.

Exclusion criteria

1. Known severe hypersensitivity to Erlotinib any of the excipient of this product. Hypersensitivity to Capecitabine, doxifluridine, or 5-FU.
2. Other coexisting malignancies or malignancies diagnosed within the last 5 years, with the exception of basal cell carcinoma, non-invasive early stage bladder cancer (<T1), and cervical cancer in situ.
3. Uncontrolled, intercurrent illness including (but not limited to) ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, or St John's Wort. Careful monitoring of PT/INR must be done for patients taking Warfarin.
5. Incomplete healing from previous oncologic or other major surgery.
6. Gastrointestinal tract disease resulting in an inability to take oral medication.
7. Pregnant women are excluded from this study because Erlotinib is an epidermal growth factor inhibitor with the potential for teratogenic or abortifacient effects based on the data suggesting that EGFR expression is important for normal organ development. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Erlotinib, breastfeeding should be discontinued if the mother is treated with Erlotinib. Capecitabine is also potentially teratogenic and its metabolites can be found in breast milk.
8. Patients with known AIDS or who are HIV-positive on anti-retroviral therapy are excluded since patients' immune deficiency are at increased risk of lethal infection when treated with marrow-suppressive therapy, and interactions between Erlotinib and anti-retroviral therapy are unknown. If patients have known risk factors of HIV they should be tested based on the discretion of the treating oncologist.
9. Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded).
10. Previous radiation to the abdomen.
11. Previous chemotherapy for pancreatic cancer.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-03-16 (Actual); Primary Completion 2013-12-27 (Actual); Study Completion 2019-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amol Narang, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not intended to be shared with other researchers, although summary of findings will be made available. In the event individual participant data is requested as support for the summary data, this data will be made available following confirmation that all patient identifiers have been "de-identified"

REFERENCES:
- [Result] Herman JM, Fan KY, Wild AT, Hacker-Prietz A, Wood LD, Blackford AL, Ellsworth S, Zheng L, Le DT, De Jesus-Acosta A, Hidalgo M, Donehower RC, Schulick RD, Edil BH, Choti MA, Hruban RH, Pawlik TM, Cameron JL, Laheru DA, Wolfgang CL. Phase 2 study of erlotinib combined with adjuvant chemoradiation and chemotherapy in patients with resectable pancreatic cancer. Int J Radiat Oncol Biol Phys. 2013 Jul 15;86(4):678-85. doi: 10.1016/j.ijrobp.2013.03.032. PMID 23773391
- See also: clinicaltrials.gov — https://clinicaltrials.gov/ct2/show/NCT00962520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients enrolled at Johns Hopkins
Groups:
- Erlotinib and EBRT After Pancreatectomy: Patients received intensity modulated radiation therapy given concurrently with erlotinib and capecitabine.
Period: Overall Study
Arm/Group | Erlotinib and EBRT After Pancreatectomy
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Erlotinib and EBRT After Pancreatectomy: All patients received RT, Erlotinib and Capecitabine, followed by gemcitabine/erlotinib
Arm/Group | Erlotinib and EBRT After Pancreatectomy
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 18
Age, Continuous [Median (Full Range); unit: years] | 62 [40 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 41
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Free Survival
Description: Time from surgery to recurrence
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Erlotinib and EBRT After Pancreatectomy: Patients received intensity modulated radiation therapy given concurrently with erlotinib and capecitabine, followed by adjuvant chemotherapy with gemcitabine/erlotinib.
Arm/Group | Erlotinib and EBRT After Pancreatectomy
Number analyzed (Participants) | 48
months | 15.6 [13.4 to 17.9]

2. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of participants experiencing adverse events during chemoradiation and during adjuvant chemotherapy, Grade 2 or higher, as defined by National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0. This is used to determine the Toxicity profile.
Time Frame: up to 3 years
Population: 39/48 total participants received maintenance chemotherapy after chemoradiation.
Measure: Count of Participants; unit: Participants
Groups:
- Chemoradiation Plus Erlotinib: Adjuvant treatment with erlotinib 100 mg plus Capecitabine 800 mg/m2 PO BID (5 days on/ 2 days off regimen) and External Beam Radiation Therapy (EBRT) at doses of 50.4 Gy in 28 fractions after pancreatectomy (Dosing for capecitabine and erlotinib was amended after considering the toxicity profile of the first 6 patients).
  erlotinib hydrochloride: Erlotinib 100 mg PO QD (1 hour prior to Capecitabine) (both given daily without interruption)
- Adjuvant Gemcitabine Plus Erlotinib: Approximately 4-8 weeks after the conclusion of chemoradiation, it is recommended patients will continue treatment with 4 cycles of gemcitabine 1000 mg/m2 days 1, 8, and 15 every 28 days plus daily erlotinib 100 mg.
Arm/Group | Chemoradiation Plus Erlotinib | Adjuvant Gemcitabine Plus Erlotinib
Number analyzed (Participants) | 48 | 39
Participants
  Grade 2 | 24 | 15
  Grade 3 | 15 | 14
  Grade 4 | 1 | 3

3. Secondary Outcome: Change in Quality of Life (QoL) as Assessed by EORTC QLQ-C30 (Version 3.0)
Description: Quality of life (QOL) was assessed before chemoradiation therapy (CRT) was started or during the first week of its administration [baseline (BL)], between completion of CRT and starting maintenance chemotherapy [time 1 (t1)], and within 3 months after completion of maintenance chemotherapy [time 2 (t2)]. European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) assesses quality of life on three domains: symptoms (score ranges from 7-14); function (score range 21-82); and global health status (score range 2-14). Higher or increasing scores mean worse outcomes; lower or decreasing scores mean better outcomes.
Time Frame: Up to 3 months after completion of maintenance chemotherapy
Population: QoL data was only available for 33 participants. Paired data for time 1 was only available for 30/33 participants, and only 20/33 participants at time 2.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Erlotinib and EBRT After Pancreatectomy
Number analyzed (Participants) | 33
score on a scale
  Global (Time 1 vs. BL): number analyzed (Participants) | 30
  Global (Time 1 vs. BL) | 1 [-6.5 to 8.5]
  Global (Time 2 vs. BL): number analyzed (Participants) | 20
  Global (Time 2 vs. BL) | -1.8 [-8.1 to 4.5]
  Global (Time 2 vs. Time 1): number analyzed (Participants) | 20
  Global (Time 2 vs. Time 1) | 4.6 [-3.3 to 12.6]
  Functional (F) - Physical (Time 1 vs. BL): number analyzed (Participants) | 30
  Functional (F) - Physical (Time 1 vs. BL) | 0.5 [-4.8 to 5.8]
  F - Physical (Time 2 vs. BL): number analyzed (Participants) | 20
  F - Physical (Time 2 vs. BL) | -3.2 [-8.8 to 2.3]
  F - Physical (Time 2 vs. Time 1): number analyzed (Participants) | 20
  F - Physical (Time 2 vs. Time 1) | -6.2 [-11 to 1.5]
  F - Role (Time 1 vs. BL): number analyzed (Participants) | 30
  F - Role (Time 1 vs. BL) | -3.1 [-13.5 to 7.2]
  F - Role (Time 2 vs. BL): number analyzed (Participants) | 20
  F - Role (Time 2 vs. BL) | -0.3 [-13.5 to 12.9]
  F - Role (Time 2 vs. Time 1): number analyzed (Participants) | 20
  F - Role (Time 2 vs. Time 1) | -4.4 [-15.5 to 6.7]
  F - Cognition (Time 1 vs. BL): number analyzed (Participants) | 30
  F - Cognition (Time 1 vs. BL) | -2.6 [-7.4 to 2.2]
  F - Cognition (Time 2 vs. BL): number analyzed (Participants) | 20
  F - Cognition (Time 2 vs. BL) | 1.2 [-6.6 to 9.1]
  F - Cognition (Time 2 vs. Time 1): number analyzed (Participants) | 20
  F - Cognition (Time 2 vs. Time 1) | -1.2 [-8.3 to 5.8]
  F - Emotional (Time 1 vs. BL): number analyzed (Participants) | 30
  F - Emotional (Time 1 vs. BL) | -0.4 [-5.3 to 4.4]
  F - Emotional (Time 2 vs. BL): number analyzed (Participants) | 20
  F - Emotional (Time 2 vs. BL) | 2.2 [-5.2 to 9.6]
  F - Emotional (Time 2 vs. Time 1): number analyzed (Participants) | 20
  F - Emotional (Time 2 vs. Time 1) | -0.6 [-9.1 to 7.9]
  F - Social (Time 1 vs. BL): number analyzed (Participants) | 30
  F - Social (Time 1 vs. BL) | 3.9 [-5.4 to 13.1]
  F - Social (Time 2 vs. BL): number analyzed (Participants) | 20
  F - Social (Time 2 vs. BL) | 4.4 [-5.7 to 14.5]
  F - Social (Time 2 vs. Time 1): number analyzed (Participants) | 20
  F - Social (Time 2 vs. Time 1) | -3.8 [-14.2 to 6.7]
  Financial (Time 1 vs. BL): number analyzed (Participants) | 30
  Financial (Time 1 vs. BL) | 1.7 [-4.3 to 7.6]
  Financial (Time 2 vs. BL): number analyzed (Participants) | 20
  Financial (Time 2 vs. BL) | 2.5 [-2.7 to 7.7]
  Financial (Time 2 vs. Time 1): number analyzed (Participants) | 20
  Financial (Time 2 vs. Time 1) | 0 [-7.6 to 7.6]
  General Symptoms (GS) - Fatigue (Time 1 vs. BL): number analyzed (Participants) | 30
  General Symptoms (GS) - Fatigue (Time 1 vs. BL) | 5.7 [-1.1 to 12.4]
  GS - Fatigue (Time 2 vs. BL): number analyzed (Participants) | 20
  GS - Fatigue (Time 2 vs. BL) | 5.2 [-2.1 to 12.5]
  GS - Fatigue (Time 2 vs. Time 1): number analyzed (Participants) | 20
  GS - Fatigue (Time 2 vs. Time 1) | 1.7 [-6.2 to 9.5]
  GS - Nausea/Vomiting (Time 1 vs. BL): number analyzed (Participants) | 30
  GS - Nausea/Vomiting (Time 1 vs. BL) | 2.5 [-2.9 to 7.9]
  GS - Nausea/Vomiting (Time 2 vs. BL): number analyzed (Participants) | 20
  GS - Nausea/Vomiting (Time 2 vs. BL) | 0 [-7.4 to 7.4]
  GS - Nausea/Vomiting (Time 2 vs. Time 1): number analyzed (Participants) | 20
  GS - Nausea/Vomiting (Time 2 vs. Time 1) | 1.9 [-5.3 to 9]
  GS - Pain (Time 1 vs. BL): number analyzed (Participants) | 30
  GS - Pain (Time 1 vs. BL) | 2.7 [-4.9 to 10.3]
  GS - Pain (Time 2 vs. BL): number analyzed (Participants) | 20
  GS - Pain (Time 2 vs. BL) | 7.2 [-2 to 16.4]
  GS - Pain (Time 2 vs. Time 1): number analyzed (Participants) | 20
  GS - Pain (Time 2 vs. Time 1) | 5 [-4 to 14]
  GS - Dyspnea (Time 1 vs. BL): number analyzed (Participants) | 30
  GS - Dyspnea (Time 1 vs. BL) | 1.7 [1.7 to 5.1]
  GS - Dyspnea Time 2 vs. BL): number analyzed (Participants) | 20
  GS - Dyspnea Time 2 vs. BL) | 3.8 [-5 to 12.5]
  GS - Dyspnea (Time 2 vs. Time 1): number analyzed (Participants) | 20
  GS - Dyspnea (Time 2 vs. Time 1) | 1.2 [-7.6 to 10.1]
  GS - Insomnia (Time 1 vs. BL): number analyzed (Participants) | 30
  GS - Insomnia (Time 1 vs. BL) | -2.5 [-9.6 to 4.6]
  GS - Insomnia (Time 2 vs. BL): number analyzed (Participants) | 20
  GS - Insomnia (Time 2 vs. BL) | 0 [-13.2 to 13.2]
  GS - Insomnia (Time 2 vs. Time 1): number analyzed (Participants) | 20
  GS - Insomnia (Time 2 vs. Time 1) | 2.5 [-8.8 to 13.8]
  GS - Appetite Loss (Time 1 vs. BL): number analyzed (Participants) | 30
  GS - Appetite Loss (Time 1 vs. BL) | -2.5 [-11.5 to 6.5]
  GS - Appetite Loss (Time 2 vs. BL): number analyzed (Participants) | 20
  GS - Appetite Loss (Time 2 vs. BL) | -15 [-28.9 to 1.1]
  GS - Appetite Loss (Time 2 vs. Time 1): number analyzed (Participants) | 20
  GS - Appetite Loss (Time 2 vs. Time 1) | -5 [-18.5 to 8.5]
  GS - Constipation (Time 1 vs. BL): number analyzed (Participants) | 30
  GS - Constipation (Time 1 vs. BL) | -4.2 [-10.7 to 2.4]
  GS - Constipation (Time 2 vs. BL): number analyzed (Participants) | 20
  GS - Constipation (Time 2 vs. BL) | -2.5 [-7.7 to 2.7]
  GS - Constipation (Time 2 vs. Time 1): number analyzed (Participants) | 20
  GS - Constipation (Time 2 vs. Time 1) | 0 [-5.4 to 5.4]
  GS - Diarrhea (Time 1 vs. BL): number analyzed (Participants) | 30
  GS - Diarrhea (Time 1 vs. BL) | 14.7 [6.8 to 22.5]
  GS - Diarrhea (Time 2 vs. BL): number analyzed (Participants) | 20
  GS - Diarrhea (Time 2 vs. BL) | 8.8 [0 to 17.5]
  GS - Diarrhea (Time 2 vs. Time 1): number analyzed (Participants) | 20
  GS - Diarrhea (Time 2 vs. Time 1) | -6.2 [-16.9 to 4.4]

4. Secondary Outcome: Change in QoL as Assessed by QLQ-PAN 26
Description: Quality of life (QOL) was assessed before CRT was started or during the first week of its administration (baseline [BL]), between completion of CRT and starting maintenance chemotherapy (time 1 [t1]), and within 3 months after completion of maintenance chemotherapy (time 2 [t2]). QLQ-PAN 26 questionnaire includes 26 questions, organized into 7 scales, with scores for each ranging from 0-100. Higher scores indicate worse health state. Therefore, decreasing (negative) scores indicate a better outcome.
Time Frame: 3 months
Population: as for outcome 3
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Erlotinib and EBRT After Pancreatectomy
Number analyzed (Participants) | 33
score on a scale
  Pancreatic Pain (t1 vs. BL): number analyzed (Participants) | 30
  Pancreatic Pain (t1 vs. BL) | -1.9 [-6.8 to 3]
  Pancreatic Pain (t2 vs. BL): number analyzed (Participants) | 20
  Pancreatic Pain (t2 vs. BL) | -3.8 [-11.7 to 4.1]
  Pancreatic Pain (t2 vs. t1): number analyzed (Participants) | 20
  Pancreatic Pain (t2 vs. t1) | 2.4 [-4.3 to 9.2]
  Digestive (t1 vs. BL): number analyzed (Participants) | 30
  Digestive (t1 vs. BL) | -0.9 [-9.1 to 7.3]
  Digestive (t2 vs. BL): number analyzed (Participants) | 20
  Digestive (t2 vs. BL) | -4.6 [-13.6 to 4.4]
  Digestive (t2 vs. t1): number analyzed (Participants) | 20
  Digestive (t2 vs. t1) | -1.4 [-7.4 to 4.6]
  Altered Bowel Habits (t1 vs. BL): number analyzed (Participants) | 30
  Altered Bowel Habits (t1 vs. BL) | 14.7 [6 to 23.5]
  Altered Bowel Habits (t2 vs. BL): number analyzed (Participants) | 20
  Altered Bowel Habits (t2 vs. BL) | 7.2 [-2.7 to 17.1]
  Altered Bowel Habits (t2 vs. t1): number analyzed (Participants) | 20
  Altered Bowel Habits (t2 vs. t1) | -4.9 [-12 to 2.3]
  Jaundice (t1 vs. BL): number analyzed (Participants) | 30
  Jaundice (t1 vs. BL) | -1.3 [-6.7 to 4]
  Jaundice (t2 vs. BL): number analyzed (Participants) | 20
  Jaundice (t2 vs. BL) | -2 [-12.1 to 8.1]
  Jaundice (t2 vs. t1): number analyzed (Participants) | 20
  Jaundice (t2 vs. t1) | 0 [-5.2 to 5.2]
  Body Image (t1 vs. BL): number analyzed (Participants) | 30
  Body Image (t1 vs. BL) | -6.2 [-13.2 to 0.7]
  Body Image (t2 vs. BL): number analyzed (Participants) | 20
  Body Image (t2 vs. BL) | -3.1 [-10.7 to 4.4]
  Body Image (t2 vs. t1): number analyzed (Participants) | 20
  Body Image (t2 vs. t1) | -0.7 [-10.2 to 8.9]
  Satisfaction with healthcare (t1 vs. BL): number analyzed (Participants) | 30
  Satisfaction with healthcare (t1 vs. BL) | 4.1 [-5.8 to 13.9]
  Satisfaction with health care (t2 vs. BL): number analyzed (Participants) | 20
  Satisfaction with health care (t2 vs. BL) | 3.1 [-12.3 to 18.5]
  Satisfaction with health care (t2 vs. t1): number analyzed (Participants) | 20
  Satisfaction with health care (t2 vs. t1) | 0 [-11.4 to 11.4]
  Sexual function (t1 vs. BL): number analyzed (Participants) | 30
  Sexual function (t1 vs. BL) | -0.5 [-10.8 to 9.7]
  Sexual function (t2 vs. BL): number analyzed (Participants) | 20
  Sexual function (t2 vs. BL) | 14.7 [2.6 to 26.8]
  Sexual function (t2 vs. t1): number analyzed (Participants) | 20
  Sexual function (t2 vs. t1) | 14.1 [3 to 25.2]

5. Secondary Outcome: Time to Death as Assessed by Median Overall Survival (Months)
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Erlotinib and EBRT After Pancreatectomy: Adjuvant treatment with erlotinib 100 mg plus Capecitabine 800 mg/m2 PO BID (5 days on/ 2 days off regimen) and External Beam Radiation Therapy (EBRT) at doses of 50.4 Gy in 28 fractions after pancreatectomy (Dosing for capecitabine and erlotinib was amended after considering the toxicity profile of the first 6 patients).
  Approximately 4-8 weeks after the conclusion of chemoradiation, it is recommended patients will continue treatment with 4 cycles of gemcitabine 1000 mg/m2 days 1, 8, and 15 every 28 days plus daily erlotinib 100 mg.
  erlotinib hydrochloride: Erlotinib 100 mg PO QD (1 hour prior to Capecitabine) (both given daily without interruption)
Arm/Group | Erlotinib and EBRT After Pancreatectomy
Number analyzed (Participants) | 48
months | 24.39 [18.87 to 29.65]

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected for approximately 3 years.
Groups:
- Erlotinib and EBRT After Prostatectomy: Patients receive oral erlotinib hydrochloride once a day for 3-5 days. Patients then proceed to surgery.
  erlotinib hydrochloride: Given orally
Arm/Group | Erlotinib and EBRT After Prostatectomy
All-Cause Mortality (participants affected / at risk) | 20/48
Serious Adverse Events (participants affected / at risk) | 16/48
Other Adverse Events (participants affected / at risk) | 31/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib and EBRT After Prostatectomy (N=48)
Fever (General disorders) | 4
Gastrointestinal bleeding (Blood and lymphatic system disorders) | 3
Altered Mental Status (Psychiatric disorders) | 2
Syncope (Nervous system disorders) | 2
Small bowel obstruction (Gastrointestinal disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Intractable nausea/vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib and EBRT After Prostatectomy (N=48)
Elevated AST/elevated ALT (Blood and lymphatic system disorders) | 12
Elevated ALP (Blood and lymphatic system disorders) | 7
Hyperbilirubinemia (Hepatobiliary disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 8
Nausea (General disorders) | 31
Dermatitis (Skin and subcutaneous tissue disorders) | 28
Anorexia (General disorders) | 30
Fatigue (General disorders) | 29
Weight loss (General disorders) | 29
Neutropenia (Blood and lymphatic system disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT00313560/Prot_SAP_000.pdf